# Title:

# RELATION BETWEEN MUSCLE FATIGUE AND TIME USE OF SMARTPHONE IN SCHOOL AGE CHILDREN

NCT: not yet assigned

Document Date: 12/11/2019

# FACULTY OF PHYSICAL THERAPY APPLICATION FOR ETHICAL REVIEW

# **NOTES:**

- Answers to questions must be entered in the space provided.
- If you have any queries about the form, please address them to the Research Ethics Team
  .

# FACULTY OF PHYSICAL THERAPY APPLICATION FOR ETHICAL REVIEW

OFFICE USE ONLY:
Application No:
Date Received:

# 1. TITLE OF PROPOSAL

# RELATION BETWEEN MUSCLE FATIGUE AND TIME USE OF SMARTPHONE IN SCHOOL AGE CHILDREN

| 2. THIS PROPOSAL IS: | |
|---|---|
| Physical Therapy Staff Research <b>Proposal</b> | |
| Physical Therapy Postgraduate Research (PGR <b>⊤\$</b> tudent Proposal √ ☐ | |
| Ma | aster □ Doctoral √ □ Other □ |
| Other Please specify): | |
| 3. INVESTIGATORS | |
| a) PLEASE GIVE DETAILS OF Studen | nt (FOR PGR STUDENT PROPOSAL) or first author |
| for staff Research Proposal | |
| Name: Title / first name / family name | Rana nabil hussien |
| Highest qualification & position held: | MSc. Of Pediatric Physical Therapy, Assistant Lecturer at MTI University |
| Department/ Faculty/ University Telephone: | Pediatrics/Physical Therapy/MTI university |
| Email address: | +2 01061164676 |
| | Rozo_elagouz25 @yahoo.com |
| a) PLEASE GIVE DETAILS OF ANY CO-SUPERVISORS OR CO-INVESTIGATORS (FOR PGR STUDENT PROPOSAL) or co- first author for staff Research Proposal b) | |
| Name: Title / first name / family name | Prof. AMIRA EL-TOHAMY |
| Highest qualification & position held: Department/ Faculty/ University | Professor |
| Telephone: | Pediatrics/Physical Therapy/ Cairo University |
| Email address: | |
| | amiraeltahamy@yahoo.com |
| Nome: Tills (first areas (first)) | DR. MOHAMED HAMED RASHAD |
| Name: Title / first name / family name Highest qualification & position held: | |
| Department/ Faculty/ University | Lecturer of Neurology Podiatrice/Medicine/ Coiro University |
| Telephone:<br>Email address: | Pediatrics/Medicine/ Cairo University |
| Lindii dudicəs. | |

# 4. SUMMARY OF PROPOSAL

To investigate the electrical muscle activity during used mobile phone

## **PURPOSE:**

- To investigate the electrical muscle activity during used mobile phone
- To investigate the most durable time to use smart phone
- To avoid development of abnormal posture by used smart phone

# **BACKGROUND:**

Using a smart phone while adopting a poor posture can cause various physical problems. The neck and shoulders are particularly vulnerable to pain due to smart phone use, with the muscles showing a high level of muscle fatigue, resulting in exhaustion and pain, Therefore, determining the durable time to use the smart phone will protect us from abnormal posture and protect our muscle and ligaments.

Furthermore avoid the incorrect position of use smartphone position.

#### **HYPOTHESES:**

- There are no statistical significant relation between time of used smart phone and muscle fatigue.

# **RESEARCH QUESTION:**

Is there a relation between time use of smart phone and muscle fatigue?

# 5. CONDUCT OF PROJECT

Please give a description of the research methodology that will be used

| 1-Electromyography (EMG) will be used to measure mean square (RMS) and maximum volu | untary |
|---|---|
| isometric contraction (MVIC) | |

# 6. PARTICIPANTS AS THE SUBJECTS OF THE RESEARCH

Describe the number of participants and important characteristics (such as age, gender, intellectual ability etc.). Specify any inclusion/exclusion criteria to be used.

one hundred fifty healthy children of both genders will participate in this study. Activity

Note: Attach a copy of any poster(s), advertisement(s) or letter(s) to be used for recruitment.
Inclusion criteria:

- -Inclusion criteria:
- 1. Their ages ranges from 12-14 years.
- 2. Subjects of school age childhood.
- 3. Not rolled on any regular athletic activity.
- 4. Children should be at the same socioeconomic level.
- -Exclusion criteria:
- 1.Individual with neck pain
- 2. Any upper limb and spinal deviation.
- 3. Worker children.

# 8. CONSENT

Describe the process that the investigator(s) will be using to obtain valid consent. If consent is not to be obtained explain why. If the participants are minors or for other reasons are not competent to consent, describe the proposed alternate source of consent, including any permission / information letter to be provided to the person(s) providing the consent.

| information fetter to be provided to the person(s) providing the consent. |
|---|
| I am freely and voluntarily consent to participate in a research program under the direction of M.Sc. |
| A thorough description of the procedure has been explained and I understand that I may withdraw my |
| consent and discontinue participation in this research at any time without prejudice to me. |
| Date Participant |
| Note: Attach a copy of the Consent Form, Participant Information Sheet (if applicable). |

## PARTICIPANT WITHDRAWAL

a) Describe how the participants will be informed of their right to withdraw from the project.

They can withdraw at anytime without prejudice to them as mention in signed consent.

| 1 | <ul> <li>b) Explain any consequences for the participant of withdrawing from the study and indicate what</li> <li>will be done with the participant's data if they withdraw.</li> </ul> | | | | | |
|---|---|---|---|---|---|---|
| | No consequences will take place. They have the utmost freedom. | | | | | |
| 9. | CONF | IDENTIA | ALITY | | | |
| | | a)<br>b) | | ants be anonymetreated as con | Yes √ □<br>Yes √ □ | No 🖰 |
| Note | Note: Participants' identity/data will be confidential if an assigned ID code or number is used, but it will not be anonymous. Anonymous data cannot be traced back to an individual participant. | | | | | |
| | 10. SIGNIFICANCE/BENEFITS Outline the potential significance and/or benefits of the research | | | | | |
| Delay in the treatment of extended Erb's palsy may result in substantial and chronic impairment due to many causes. One of the causes is the imbalance between the recovery of elbow lexors and elbow extensors where the latter will be delayed. This study will determine if a debilitating tightness and contracture (elbow flexion) can be prevented using the kinesiology tape in infants with Extended Erb's Palsy. | | | | | | |
| 11. RIS | sks | | | | | |
| Outline any potential risks to <b>INDIVIDUALS</b> , including research staff, research participants, other individuals not involved in the research and the measures that will be taken to | | | | | | |
| <u>,</u> | <u>minimi</u> | | any risks and | | | vent of mishap |
| Risk of Infection: minimizing the risk through adequate sterilization of the treated areas during evaluation and treatment. | | | | | | |

# 12. DECLARATION BY APPLICANTS

I submit this application on the basis that the information it contains is confidential and will be used by the Faculty of Physical Therapy for the purposes of ethical review and monitoring of the research project described herein, and to satisfy reporting requirements to regulatory bodies. The information will not be used for any other purpose without my prior consent.

# I declare that:

- The information in this form together with any accompanying information is complete and correct to the best of my knowledge and belief and I take full responsibility for it.
- I will report any changes affecting the ethical aspects of the project to the Faculty of Physical Therapy Research Ethics Officer.
- I will report any adverse or unforeseen events which occur to the relevant Ethics Committee via the Faculty of Physical Therapy Research Ethics Officer.

| Name of Principal investigator/project supervisor: | Rana nabil hussien |
|----------------------------------------------------|-----------------------|
| | Prof. Amera El-Tohamy |
| Date: | 12 of novamber, 2019 |

# **Preflight Results**

# **Document Overview**

# **Preflight Information**

Title: Profile: Convert to PDF/A-1b

Author: El Khatib, Yehia (elkhatib) Version: Qoppa jPDFPreflight v2020R2.00 Creator: Microsoft® Word 2010 Date: Sep 20, 2020 12:14:37 PM

Producer: Microsoft® Word 2010

Legend: (X) - Can NOT be fixed by PDF/A-1b conversion.

(!X) - Could be fixed by PDF/A-1b conversion. User chose to be warned in PDF/A settings.


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Bold is not embedded. Font Times New Roman, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Bold is not embedded. Font Times New Roman, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman,Bold is not embedded. Font Times New Roman,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Bold is not embedded. Font Times New Roman, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed


- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed 7 more not displayed


(X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed


- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 3 more not displayed


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Italic is not embedded. Font Times New Roman, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman, Italic is not embedded. Font Times New Roman, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed 26 more not displayed


(X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed - 51 more not displayed


- $\bar{(}X)$  Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed


- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 21 more not displayed


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed


- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 35 more not displayed


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Italic is not embedded. Font Arial, Italic can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed 7 more not displayed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 20 more not displayed


- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed


- (X) Font Arial,Bold is not embedded. Font Arial,Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Arial, Bold is not embedded. Font Arial, Bold can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Times New Roman is not embedded. Font Times New Roman can not be embedded because: Could not find matching font to embed
- (X) Font Arial is not embedded. Font Arial can not be embedded because: Could not find matching font to embed 24 more not displayed